CLINICAL TRIAL: NCT00602394
Title: A Single Dose, Two-Period, Two-Treatment Crossover Bioequivalency Study of 300 mg Lithium Carbonate Extended Release Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of 300 mg Lithium Carbonate Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LITH-12
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lithium

SUMMARY:
The objective of this study was the bioequivalence of a Roxane lithium carbonate 300 mg extended release tablet formulation compared to Solvay's Lithobid 300 mg extended release tablet under fed conditions using a single-dose, randomized, 2 treatment, 2-period, 2-sequence crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to lithium, or any comparable or similar product.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2003-05; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Fourteen day washout

CONTACTS AND LOCATIONS:
Overall Officials: So R Hong, MD, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, 11248 Wilcrest Green, , Houston77042, Houston, Texas, United States